CLINICAL TRIAL: NCT07197593
Title: Validity and Reliability of Calf Raise Tests in Patients With Achilles Tendon Rupture and Lateral Ankle Sprain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Responsible Party: Principal Investigator, Nicola Maffiuletti, Head of Research Group, Human Performance Lab, Schulthess Klinik
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2025-01043
Record Dates: First submitted 2025-09-05; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Achilles Tendon; Ankle Sprain
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Intervention Model Description: Validity and reliability study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Calf Raise Test (CRT) App (Other): The validated CRT App allows to accurately measure work, power and peak height in in individuals performing the calf raise test.
  Interventions: Other: Calf Raise Test

INTERVENTIONS:
Other: Calf Raise Test — The study participants perform three single-leg CRTs (tracked by the CRT App) in a fixed sequence: concentric power, eccentric-concentric power and endurance. ATRC/LAS Individuals start with the affected leg, healthy participants with the dominant leg.

SUMMARY:
This study aims to evaluate the validity and reliability of clinically used Calf Raise Test parameters (collected with the "the Calf Raise App") between patients with Lateral Ankle Sprain or Achilles Tendon Repair and healthy controls.

DETAILED DESCRIPTION:
Lateral ankle sprains (LAS) are the most common lower limb injury in sports, affecting the lateral ligament complex in 80% of cases. Diagnosis is based on clinical evaluation (mechanism of injury, history, weight-bearing status, ligament integrity tests) and conservative treatment is recommended in the absence of additional injuries. However, up to 40% of LAS patients develop chronic ankle instability (CAI), that is characterized by persistent pain, instability, and recurrent sprain. Despite the absence of direct injury to the calf muscle-tendon unit, LAS patients may experience plantar flexor strength deficits for up to 6 months, making calf function assessment crucial for rehabilitation and return to sport purposes. The International Ankle Consortium Rehabilitation-Oriented Assessment (ROAST) recommends isokinetic and hand-held dynamometry for muscle strength testing; however, these methods are often impractical in clinical settings. As a result, the single-leg heel raise test (calf raise test) is already widely used in clinical practice as a pragmatic alternative to assess plantar flexor function and to monitor rehabilitation progress over time.

Achilles tendon rupture (ATR) is another common injury that severely impacts calf muscle-tendon function. The Achilles tendon, formed by the gastrocnemius and soleus muscles, is the strongest tendon in the human body and can withstand forces up to 17 times body weight. Ruptures occur when the tendon is overstretched, with elongation beyond 8% resulting in visible structural failure. Recent epidemiological data point to an incidence of ATR of 41.7 cases per 100,000 person-years in Sweden and 29.3 per 100,000 person-years in Ontario, Canada, with men aged 30-50 being the most affected.

In both LAS and ATR patients, the evaluation of calf muscle-tendon function is essential for individualized rehabilitation and for monitoring functional recovery over time. The calf raise test (CRT) is a widely used tool for evaluating calf muscle-tendon function, with good validity and reliability (intraclass correlation coefficients [ICC] of 0.57 to 0.99 and Pearson's correlation coefficients [r] of 0.56 to 0.98). Traditionally, the CRT measures muscular endurance by counting repetitions until task failure. However, recent research suggests that peak displacement and power output may be more sensitive indicators of functional deficits in Achilles tendon rehabilitation. Additionally, measuring power alongside endurance may better reflect the demands of sport-related activities.

Although such parameters have long been measurable in laboratory settings, these technologies are expensive, require specialized personnel, and are often inaccessible in routine clinical environments. Recent advances in digital health technology-most notably the development of validated mobile applications such as the Calf Raise App-now enable reliable, objective, and cost-efficient quantification of displacement, power and work during the CRT. As such, calf raise power obtained during a modified app-controlled CRT has shown a significant correlation with 10-m sprint times in rugby players (R² values ranging from 0.25 to 0.39, p < 0.05).

Despite the frequent use of various CRTs in rehabilitation settings for LAS and ATR patients, several important aspects remain unexplored. Specifically:

* The discriminative (known group) validity of CRT-derived endurance to distinguish LAS patients from healthy individuals has not yet been established.
* In the same way, the discriminative validity of CRT-derived power to differentiate LAS or ATR patients from healthy controls is not known.
* The inter-tester reliability of CRT-derived endurance has not been assessed specifically in LAS patients.
* Similarly, the inter-tester reliability of CRT-derived power has never been evaluated in either LAS or ATR patients.

This study is designed to fill these gaps by systematically evaluating the discriminative validity of clinically used CRT parameters between patients with LAS or ATR and healthy controls, as well as the inter-tester reliability of these parameters within patient groups.

ELIGIBILITY:
General Inclusion Criteria:

* Signed informed consent
* Aged 18-65 years
* German or English speaking

Inclusion Criteria:

LAS individuals: Unilateral LAS 4-16 weeks post-injury diagnosed by a physician as LAS, supination trauma, ankle distortion or ligamentous ankle injury.

ATR individuals: Unilateral ATR 6- 24 months post-injury/surgery (surgical or conservative treatment).

Healthy controls: Matched to Patients by Group Level: Physical Activity, Age and Gender.

Exclusion Criteria:

LAS individuals: Medial Ligament injuries (Grade II or III) ATR individuals: Previous ATR

General Exclusion Criteria:

* Chronic Ankle Instability (defined by symptoms such as giving way, perceived instability and at least one LAS within the last 6 months)
* Previous ATR
* Other lower limb injury and/or surgery in the last year (e.g. fractures, ligament reconstructions or other conditions resulting in ≥ 6 months of sports inactivity)
* Impaired motor function of the lower limb due to neurovascular or neurological diseases
* Vestibular or visual disturbances
* Or any other pathoanatomic abnormality that would affect motor performance (e.g. foot arthrodesis, toe amputation/missing toes or other conditions such as joint deformities, severe chronic pain).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Calf Raise Test (CRT) | The CRT data will be collected at two time points: at baseline and after a 30- min break. Total time of data collection: ca. 1 hour.
  The CRT (evaluated by the use of the CRT App) yields three different variables of interest:
  * Concentric power CRT: peak power (W) during the ascending phase
  * Eccentric-concentric power CRT: peak power (W) during the ascending phase
  * Endurance CRT: number of repetitions (n), total positive work (W), and total positive displacement (cm)

SECONDARY OUTCOMES:
Patient-reported outcome measures (PROM) - FAOS | This PROM data will be collected at one time point: at baseline.
  For ATR patients, LAS patients and healthy controls _ specific score I:
  Foot and Ankle Outcome Score (FAOS). This PROM consists of specific items, which produce a unique numeric score as unit measurement (outcome measure).
Patient-reported outcome measure (PROM) - ATRS | This PROM data will be collected at one time point: at baseline.
  For ATR patients and healthy controls_ specific score II:
  Achilles Tendon Total Rupture Score (ATRS). This PROM consists of specific items, which produce a unique numeric score as unit measurement (outcome measure).
Patient-reported outcome measure (PROM) - FFI | This PROM data will be collected at one time point: at baseline.
  For LAS patients and healthy controls _ specific score III:
  Functional Foot Index (FFI). This PROM consists of specific items, which produce a unique numeric score as unit measurement (outcome measure).
Patient-reported outcome measure (PROM) - FAAM | This PROM data will be collected at one time point: at baseline.
  For LAS patients and healthy controls _ specific score IV:
  Foot and Ankle Ability Measurement (FAAM). This PROM consists of specific items, which produce a unique numeric score as unit measurement (outcome measure).
Patient-reported outcome measure (PROM) - UCLA Activity Score | This PROM data will be collected at one time point: at baseline.
  For ATR patients, LAS patients and healthy controls - generic score (Physical Activity) I: UCLA Activity Score.
  This PROM consists of specific items, which produce a unique numeric score as unit measurement (outcome measure).
Patient-reported outcome measure (PROM) - GPAQ | This PROM data will be collected at one time point: at baseline.
  For ATR patients, LAS patients and healthy controls - generic score (Physical Activity) II: Global Physical Activity Questionnaire (GPAQ).
  This PROM consists of specific items, which produce a unique numeric score as unit measurement (outcome measure).

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared. The study involves sensitive clinical data that is subject to privacy protections and institutional regulations. Ownership of the data remains with the clinic, and confidentiality requirements prevent making these data publicly available.